CLINICAL TRIAL: NCT03487237
Title: Prevalence of Pulmonary Embolism in Emergency Department Patients With Isolated Syncope
Brief Title: Prevalence of PE in ED Patients With Isolated Syncope
Acronym: PEEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K171102J
Record Dates: First submitted 2018-03-01; First posted 2018-04-03 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Syncope
Keywords: Syncope; Pulmonary embolism; emergency department; clinical decision rule
MeSH Terms: conditions — Syncope; Pulmonary Embolism; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patient (Experimental): Included patients will undergo a formal work up for pulmonary embolism: Ddimer testing, followed if positive by a computed tomography pulmonary angiogram or V/Q scan.
  Interventions: Biological: Ddimer testing

INTERVENTIONS:
Biological: Ddimer testing — Included patients will undergo a formal work up for pulmonary embolism: Ddimer testing, followed if positive by a computed tomography pulmonary angiogram or V/Q scan.

SUMMARY:
Syncope is a rapid onset, transient, loss of consciousness with a short duration. This symptom has been reported to be a specific presentation of patients with pulmonary embolism. However, the prevalence of pulmonary embolism in patients with syncope remains debated. This prospective cohort study will recruit patients presenting to the emergency department with a syncope, who will systematically undergo formal workup for pulmonary embolism. The main objective of this study is to assess the prevalence of pulmonary embolism in ED patients with syncope

DETAILED DESCRIPTION:
Syncope is a rapid onset, transient, loss of consciousness with a short duration. This symptom has been reported to be a specific presentation of patients with pulmonary embolism. However, the prevalence of pulmonary embolism in patients with syncope remains debated. This prospective cohort study will recruit patients presenting to the emergency department with a syncope, who will systematically undergo formal workup for pulmonary embolism. The main objective of this study is to assess the prevalence of pulmonary embolism in ED patients with syncope

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years visiting the Emergency Department,
* history of syncope in the past 24 hours: loss of consciousness, rapid onset, short duration (<1 min), transient, with spontaneous and rapid recovery without post event confusion
* With or without prodromes
* Without any other obvious cause
* Informed written consent
* Affiliation to a social security system (AME Excepted)

Exclusion Criteria:

- Other criteria for PE suspicion : Acute onset of dyspnea Acute severe chest pain,

* Pregnancy
* Concurrent anticoagulation treatment
* Other obvious cause of syncope : Seizure, Stroke, Traumatic brain injury , toxic intake , Atrioventricular block type 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
diagnosis of Pulmonary embolism within 72 hrs after ED visit Safety | 72 hours after ED visit
  diagnosis of Pulmonary embolism within 72 hrs after ED visit ( Ddimer testing, followed if positive by a computed tomography pulmonary angiogram or V/Q scan).

SECONDARY OUTCOMES:
Validation of usual clinical decision rules-Wells | Day 0
  Wells score:
  Clinical signs and symptoms of DVT 3 Immobilization or surgery within 4 weeks 1.5 Heart rate > 100 beats per min 1.5 Previous DVT or PE 1.5 Hemoptysis 1 Malignancy 1 Alternative diagnosis is less likely than PE 3 Low: 0-1; intermediate: 2-6; high: >6
Validation of usual clinical decision rules-Revised Geneva Score | Day 0
  Age > 65 years 1 Previous DVT or PE 3 Surgery or fracture within 1 monht 2 Active malignant condition within a year 2 Unilateral lower limb pain 3 Hemoptysis 2 Heart Rate 75 - 94 beats per min 3 >94 beats per min 5 Pain on lower limb deep venous palpation and unilateral edema 5 low: 0-3; intermediate: 4-10; high: >11
Validation of usual clinical decision rules-PERC | Day 0
  PERC:
  * Age less than 50 years
  * Heart rate less than 100 beats per minute
  * No prior history of thrombo-embolic event
  * Oxygen saturation greater than 94%
  * No trauma or surgery in the past four weeks
  * No hemoptysis
  * No exogenous estrogen intake
  * No unilateral leg swelling
Prevalence of Pulmonary Embolism among patients with cancer history. | Day 28
rate of false positive of the PERC rule | 72 hours after ED visit
  Patients with a PERC=0 ultimately diagnosed with a pulmonary embolism within 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexis Raynal, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No